CLINICAL TRIAL: NCT06082050
Title: Efficacy and Safety of Intravenous YOLT-201 for Transthyretin Amyloidosis Cardiomyopathy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: YolTech Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOLT-201_2023_IIT_01
Record Dates: First submitted 2023-09-19; First posted 2023-10-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-11

CONDITIONS: Transthyroxin Amyloidosis Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- YOLT-201 (Experimental): Infusion of YOLT-201 at Day 1， Subjects may voluntarily accept the second study drug treatment at the OBD (Optimal Biological Dose) level.
  Interventions: Drug: YOLT-201

INTERVENTIONS:
Drug: YOLT-201 — Infusion of YOLT-201 at Day 1， Subjects may voluntarily accept the second study drug treatment at the OBD (Optimal Biological Dose) level.

SUMMARY:
This study is a single-arm, open-label, single-dose escalation trial aimed at evaluating the safety and tolerability of YOLT-201 treatment in patients with Transthyretin Amyloidosis Cardiomyopathy （ATTR-CM）, as well as assessing the preliminary efficacy of subjects treated with YOLT-201.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 and ≤80 years old at the time of signing informed consent.
2. Diagnosis of transthyretin cardiac amyloidosis (ATTR-CM) based on the 2021 "Chinese Expert Consensus on the Diagnosis and Treatment of Transthyretin Cardiac Amyloidosis," the 2021 European Society of Cardiology (ESC) guidelines, and the 2023 American College of Cardiology (ACC) guidelines, including hereditary ATTR cardiac amyloidosis (ATTRv-CM) and wild-type ATTR cardiac amyloidosis (ATTRwt-CM); and relevant indicators meet the following criteria:

   2.1 New York Heart Association (NYHA) functional classification of I to III; 2.2 6-minute walk test (6-MWT) ≥ 150 meters at screening; 2.3 Echocardiogram evidence of cardiac involvement: left ventricular wall thickness (interventricular septum and/or posterior wall thickness ≥12 mm); 2.4 Brain natriuretic peptide N-terminal prohormone (NT-proBNP) < 2000 pg/mL at screening; 2.5 Receiving stable and standardized cardiovascular medication treatment.
3. Body weight must not be less than 40 kg at screening.
4. Subjects must meet the following laboratory criteria at screening:

   4.1 Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (except for Gilbert's syndrome), International Normalized Ratio (INR) < upper limit of normal (ULN); 4.2 Subjects with a history of Gilbert's syndrome have a total bilirubin not exceeding twice the upper limit of normal (ULN) during the screening period; 4.3 Estimated glomerular filtration rate (eGFR) > 45 mL/min/1.73m^2 at screening; 4.4 Platelet count ≥ 100 × 10^9/L; 4.5 Coagulation function at screening: fibrinogen, activated partial thromboplastin time (APTT), prothrombin time (PT), and thrombin time (TT) are all within the normal range; 4.6 Low-density lipoprotein (LDL) cholesterol < 200 mg/dL; 4.7 Vitamin A level ≥ lower limit of normal (LLN); 4.8 Vitamin B12 level ≥ lower limit of normal (LLN).
5. Acceptance of ATTR-CM medication treatment:

   5.1 Unable to receive existing ATTR-CM-related medication due to regional medical resources, health policies, personal financial capacity, or drug intolerance; 5.2 Despite receiving at least 6 months of ATTR-CM medication treatment, the subject's ATTR-CM condition still progresses (meeting at least one of the following): Increased hospitalizations related to heart failure; Worsening of NYHA classification; 6-MWT decrease of at least 30 meters; NT-proBNP increase by 30%; Troponin increase by 30%; Echocardiogram indicates: increase in left ventricular wall thickness by 2 mm, or decrease in left ventricular ejection fraction by ≥5%, or decrease in global longitudinal strain by ≥1%, or decrease in stroke volume by ≥5%, or worsening diastolic function; New conduction block on electrocardiogram.
6. No intake of alcohol from the start of the screening period to 28 days after receiving the trial treatment medication.
7. Female subjects must be postmenopausal for at least one year, or have undergone hysterectomy.
8. Male subjects and their partners must use highly effective contraceptive measures recognized by the doctor throughout the trial process and for at least 5 months after the trial ends.
9. Male subjects must not donate sperm within 84 days after receiving study medication.
10. Voluntary signing of informed consent.

Exclusion Criteria:

1. Amyloidosis that is not related to TTR protein degeneration, such as immunoglobulin light chain (AL) amyloidosis.
2. History of multiple myeloma.
3. Indeterminate monoclonal gammopathy (MGUS) and/or immunoglobulin free light chain (FLC) ratio alterations, unless fat, bone marrow, or cardiac biopsy confirms the absence of light chains but presence of TTR protein through mass spectrometry or immunoelectron microscopy. For chronic kidney disease (CKD) subjects with no monoclonal protein in blood and urine, the acceptable FLC ratio is 0.26 to 2.25. If the risks of biopsy outweigh the benefits, different results may be discussed with local hematologists, investigators, and medical monitors.
4. Allergy to any lipid nanoparticle (LNP) components, or history of exposure to LNP components or laboratory abnormalities or adverse reaction events related to their treatment: 4.1 Normal baseline, ALT or AST > 3 × ULN or appearance of baseline triple value after receiving LNP product. 4.2 Normal baseline, INR, APTT, or D-dimer > 1.5 × ULN; if baseline is higher than normal after receiving LNP product, it is 1.5 times the baseline value. 4.3 Any adverse reactions related to LNP product treatment are defined as grade 3 or higher (CTCAE). Injection site reactions (IRR) requiring treatment or discontinuation of infusion; slowing down the infusion rate to alleviate infusion-related reactions. The investigator believes that any adverse reaction events related to LNP treatment should be excluded.
5. Use of any of the following ATTR treatments within a certain period:

   5.1 Patisiran (LNP small interfering RNA siRNA) treatment product (within 90 days after administration).

   5.2 Previous treatment with Inotersen (antisense oligonucleotide ASO) (within 160 days after administration).

   5.3 Previous use of Vutrisiran (investigational siRNA therapeutic GalNAc conjugate).

   5.4 Tafamidis (TTR stabilizer): less than 10 days since last drug administration before study drug administration.

   5.5 Diflunisal (TTR stabilizer): less than 3 days since last drug administration before study drug administration.

   5.6 Doxycycline and/or tauroursodeoxycholic acid (TTR chaperone): less than 14 days since last drug administration before study drug administration.

   5.7 Any other drugs used for the treatment of ATTR-CM: less than 30 days or 5 half-lives (whichever is longer) since last drug administration before study drug administration.
6. Other organic heart diseases, such as ischemic heart disease, uncontrolled hypertension, valvular heart disease, etc., leading to cardiomyopathy.
7. Current or previous NYHA class IV symptoms or worsening heart failure symptoms within 90 days before or during screening.
8. Hospitalization or invasive surgery due to cardiovascular and cerebrovascular diseases within 90 days before or during screening. For example, acute coronary syndrome, unstable angina, stroke, TIA, coronary artery reconstruction, cardiac device implantation, valvular repair, or major surgery, etc.
9. Expected to undergo invasive cardiovascular surgery (such as coronary artery stent, pacemaker implantation, etc.) within 28 days after medication.
10. Subjects who cannot or are unwilling to supplement vitamin A.
11. Subjects who cannot or are unwilling to accept the required medication treatment plan before treatment.
12. Antiplatelet (such as aspirin, clopidogrel) or antithrombotic treatment (such as warfarin, dabigatran, apixaban) within 14 days before study drug administration.
13. History of bleeding diathesis or coagulation disorders (such as liver cirrhosis, malignant hematological diseases, antiphospholipid antibody syndrome).
14. The investigator believes that the expected survival is less than 2 years.
15. Ophthalmological examination results consistent with vitamin A deficiency.
16. Known or suspected systemic viral, parasitic, or fungal infections, or expected to receive antibiotic treatment for bacterial infections within 14 days after screening.
17. History of hepatitis B or C infection or positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) at screening.
18. History of human immunodeficiency virus (HIV) positivity.
19. Clinically significant thyroid function abnormalities judged by the investigator.
20. History of liver, heart, or other solid organ transplantation or bone marrow transplantation within 1 year at screening, or expected transplantation. Note: No history or plan for corneal transplantation.
21. History of active malignant tumors within 5 years before screening, except for basal cell carcinoma of the skin, cured squamous cell carcinoma of the skin, cured cervical cancer, or low-grade prostate cancer under observation.
22. History of alcohol abuse or drug abuse within 3 years before screening.
23. Female subjects with childbearing potential or who are breastfeeding.
24. Other physical, social, or psychological diseases, including the use of illicit drugs or alcohol, which the investigator believes may adversely affect the subject's safety, impair the assessment of study results, or prevent the subject from complying with any conditions of this study, laboratory abnormalities, or other reasons.
25. Unwilling to comply with study procedures, including follow-ups as specified in the protocol, or unwilling to cooperate fully with the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Adverse event Adverse event Adverse events | hrough study completion, an average of 1 year
  Adverse events

SECONDARY OUTCOMES:
Cmax | hrough study completion, an average of 1 year
  Cmax
Tmax | hrough study completion, an average of 1 year
  Tmax
AUCinf | through study completion, an average of 1 year
  AUCinf
AUClast | through study completion, an average of 1 year
  AUClast
t1/2 | through study completion, an average of 1 year
  t1/2
CL/F | through study completion, an average of 1 year
  CL/F
change of TTR | through study completion, an average of 1 year
  change of TTR
change of QOL-DN | Week3,Week24,Week52
  change of QOL-DN
change of EQ-5D-5L | Week 24、Week 52
  change of EQ-5D-5L
change of 10-MWT | Week 24、Week 52
  change of 10-MWT
change of NFL | Week 3、Week 24、Week 52
  change of NFL
change of mBMI | Week 3、Week 24、Week 52
  change of mBMI
change of NT-proBNP | Week 24、Week 36、Week 52
  NT-proBNP
change of troponin | Week 24、Week 36、Week 52
  change of troponin
change of 6-MWT | Week 36、Week 52
  change of 6-MWT
change of NYHA cardiac function classification change of NYHA cardiac function classification | Week 24、Week 36、Week 52
  change of NYHA cardiac function classification NYHA cardiac function classification change of NYHA cardiac function classification
change of KCCQ | Week 24、Week 36、Week 52
  change of KCCQ
change of Interventricular septal wall thickness | Week 52
  change of Interventricular septal wall thickness on echocardiography
change of Left ventricular (LV) posterior wall thickness | Week 52
  change of Left ventricular (LV) posterior wall thickness on echocardiography
change of LV mass | Week 52
  change of LV mass on echocardiography
change of LV end-diastolic volume | Week 52
  change of LV end-diastolic volume on echocardiography
change of LV end-systolic volume | Week 52
  change of LV end-systolic volume on echocardiography
change of LV ejection fraction | Week 52
  change of LV ejection fraction on echocardiography
change of Cardiac output | Week 52
  change of Cardiac output on echocardiography
change of Global longitudinal strain | Week 52
  change of Global longitudinal strain on echocardiography
change of Left atrial size | Week 52
  change of Left atrial size on echocardiography
change of Left ventricular end-diastolic volume on Cardiac magnetic resonance | W52
  change of Left ventricular end-diastolic volume on Cardiac magnetic resonance
change of Left ventricular end-systolic volume on Cardiac magnetic resonance | Week 52
  change of Left ventricular end-systolic volume on Cardiac magnetic resonance
change of Left ventricular systolic volume on Cardiac magnetic resonance | Week 52
  change of Left ventricular systolic volume on Cardiac magnetic resonance
change of Left ventricular ejection fraction on Cardiac magnetic resonance | Week 52
  change of Left ventricular ejection fraction on Cardiac magnetic resonance
change of Overall longitudinal strain of left ventricle on Cardiac magnetic resonance | Week 52
  change of Overall longitudinal strain of left ventricle on Cardiac magnetic resonance
change of Mitral ring plane contraction displacement on Cardiac magnetic resonance | Week 52
  change of Mitral ring plane contraction displacement on Cardiac magnetic resonance
change of Left ventricular myocardial mass on Cardiac magnetic resonance | Week 52
  change of Left ventricular myocardial mass on Cardiac magnetic resonance
change of Right ventricular end-diastolic volume on Cardiac magnetic resonance | Week 52
  change of Right ventricular end-diastolic volume on Cardiac magnetic resonance
change of Right ventricular end-systolic volume on Cardiac magnetic resonance | Week 52
  change of Right ventricular end-systolic volume on Cardiac magnetic resonance
change of Right ventricular systolic volume on Cardiac magnetic resonance | Week 52
  change of Right ventricular systolic volume on Cardiac magnetic resonance
change of Right ventricular ejection fraction on Cardiac magnetic resonance | Week 52
  change of Right ventricular ejection fraction on Cardiac magnetic resonance
change of Tricuspid ring plane contraction offset on Cardiac magnetic resonance | Week 52
  change of Tricuspid ring plane contraction offset on Cardiac magnetic resonance
change of Right ventricular longitudinal strain on Cardiac magnetic resonance | Week 52
  change of Right ventricular longitudinal strain on Cardiac magnetic resonance
change of Left atrial volume on Cardiac magnetic resonance | Week 52
  change of Left atrial volume on Cardiac magnetic resonance
change of Right atrial volume on Cardiac magnetic resonance | Week 52
  change of Right atrial volume on Cardiac magnetic resonance
change of Extracellular volume on Cardiac magnetic resonance | Week 52
  change of Extracellular volume on Cardiac magnetic resonance
level of anti-drug antibody | through study completion, an average of 1 year
  level of anti-drug antibody
level of cas9 antibody | through study completion, an average of 1 year
  level of cas9 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No